CLINICAL TRIAL: NCT04430842
Title: A Phase 1, Open Label, Multi-Center, Single and Multiple Dose, Dose Escalation and Expansion Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of QBS10072S in Previously Treated Patients With Advanced or Metastatic Cancers With High LAT1 Signatures, and in Patients With Relapsed or Refractory Grade 4 Astrocytoma
Brief Title: Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of QBS10072S
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quadriga Biosciences, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QBS-72S-1001
Record Dates: First submitted 2020-06-02; First posted 2020-06-12 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Astrocytoma; Brain Cancer; Brain Metastases; Bladder Cancer; Breast Cancer; Cervical Cancer; Cholangiocarcinoma; Colorectal Cancer; Esophagus Cancer; Gastric Cancer; Head and Neck Cancer; Kidney Cancer; Liver Cancer; Lung Cancer; Melanoma; Ovarian Cancer; Pancreatic Cancer; Pleural Mesothelioma; Prostate Cancer; Sarcoma; Tongue Cancer; Thymic Carcinoma; Urinary Tract Cancer
Keywords: Phase 1; Dose escalation; Metastatic; Brain metastasis; Brain metastases; GBM; Astrocytoma; Brain tumor; Cancer; Oncology; Glioblastoma; Glioblastoma multiforme; Brain; Neurology; Neuroscience; Headaches; Vomiting; Seizures; Drowsiness; Chemotherapy; Surgery; Radiation; Neuro-oncology; Blurred vision; Loss of appetite; Speech difficulty; Changes in ability to think and learn; Changes in mood and personality; Persistent headaches; Neuropathologist; Magnetic resonance spectroscopy (MRS); Positron emission tomography (PET scan); Intraoperative MRI; Tumor removal; Craniotomy; Standard external beam radiation therapy; Radiosurgery; Temozolomide; Bevacizumab; Avastin; Neurological exam; TMZ
MeSH Terms: conditions — Astrocytoma; Brain Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Cholangiocarcinoma; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Liver Neoplasms; Lung Neoplasms; Melanoma; Ovarian Neoplasms; Pancreatic Neoplasms; Mesothelioma, Malignant; Prostatic Neoplasms; Sarcoma; Tongue Neoplasms; Thymoma; Urologic Neoplasms; Neoplasm Metastasis; Neoplasms; Glioblastoma; Headache; Vomiting; Seizures; Sleepiness; Anorexia; Speech Disorders

STUDY DESIGN:
Intervention Model Description: The dose escalation scheme for this trial employs an mTPI-2 design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation of QBS10072S (Experimental): Intravenous administration of QBS10072S once every 4 weeks starting at 3mg/m2 and increasing dose levels in subsequent cohorts.
  Interventions: Drug: QBS10072S

INTERVENTIONS:
Drug: QBS10072S — QBS10072S targets cancers with high LAT1 expression.

SUMMARY:
This is a multi-center, open-label, dose escalation study to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, and maximum tolerated dose (MTD) of QBS10072S in patients with advanced or metastatic cancers with high LAT1 expression. The MTD of QBS10072S will be confirmed in patients with relapsed or refractory grade 4 astrocytoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged ≥18 years at the time of informed consent.
2. Adequate Bone Marrow Function
3. Adequate renal function
4. Adequate Liver Function
5. Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1 except for AEs not constituting a safety risk by Investigator judgment.
6. A histological or cytological diagnosis of a solid tumor that is advanced/metastatic, patients intolerant to standard treatment or, resistant to standard therapy* (per NCCN guidelines) or for which no curative therapy is available for the following tumor types:

   - Bladder, Brain, Breast, Cervical, Cholangiocarcinoma, Colorectal, Esophageal, Gastric, Head and Neck, Kidney, Liver, Lung, Melanoma, Ovarian, Pancreatic, Pleural mesothelioma, Prostate, Sarcoma, Tongue cancer, Thymic carcinomas, Urinary tract
7. At least one measurable lesion (as defined by RECIST version 1.1) that has not been previously irradiated.
8. An ECOG PS 0 to 2.

Exclusion Criteria:

1. Patients with tumor primarily localized to the brainstem or spinal cord. Presence of known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth.
2. Patients with advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term (including patients with massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver involvement).
3. Patients with any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
4. Major surgery within 4 weeks prior to study entry.
5. Radiation therapy within 4 weeks prior to receiving the first QBS10072S dose (bone lesions requiring radiation may be treated with limited radiation therapy during this period).
6. Systemic anticancer therapy within 4 weeks prior to study entry
7. Bleeding esophageal or gastric varices <2 months prior to the date of informed consent.
8. Unmanageable ascites.
9. Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect patient safety or interpretation of study results
10. On therapeutic anticoagulation, except low molecular weight heparin, vitamin K antagonists or factor Xa inhibitors may be allowed following discussion with the Sponsor.
11. Any of the following in the previous 6 months: myocardial infarction, congenital long QT syndrome, Torsade de Pointes, clinically significant arrhythmias (including sustained ventricular tachyarrhythmia and ventricular fibrillation), left anterior hemiblock, bifascicular block, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association class III or IV), cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism or other clinical significant episode of thromboembolic disease. Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, atrial fibrillation of any grade (Grade ≥2 in the case of asymptomatic lone atrial fibrillation).
12. Hypertension that cannot be controlled by medications (>150/90 mmHg despite optimal medical therapy) or requiring more than two medications for adequate control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) | 28 days
  MTD will be determined by presence of AEs as characterized by type, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study therapy.

SECONDARY OUTCOMES:
Safety and tolerability assessed by adverse events and serious adverse events | 28 days
  Safety and tolerability will be determined by adverse events as characterized by type, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study therapy.
Peak Plasma Concentration (Cmax) | 28 days
  Determine the maximum plasma concentration of QBS10072S.
Area under the plasma concentration versus time curve (AUC) of QBS10072S | 28 days
  Determine the plasma concentration of QBS10072S over time.
Half-life of QBS10072S in plasma (t1/2) | 28 days
  Determine the half life of QBS10072S in plasma; the half-life of a drug is the time taken for the plasma concentration of a drug to reduce to half its original value.
Time to maximum concentration of QBS10072S in plasma (Tmax) | 28 days
  Determine the time it takes to achieve maximum concentration of QBS10072S in plasma.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - St George Private Hospital, Kogarah, New South Wales
  - Sydney Southwest Private Hospital, Liverpool, New South Wales